CLINICAL TRIAL: NCT02671162
Title: Evaluation the Effect of Fumaria Parviflora L. on Uremic Pruritus of End-stage Renal Disease Patients: A Randomized Double- Blind Placebo-controlled Clinical Trial
Brief Title: Evaluating the Effect of Fumaria Parviflora L. in Uremic Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Rahimeh Akrami, Dr., Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRCT2015080110410N2
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: End-Stage Renal Disease; Pruritus
Keywords: Pruritus; End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Pruritus | interventions — Flour; Fumariae herba

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wheat (Placebo Comparator): Placebo capsule/ 2 capsule 3 times per day
  Interventions: Drug: Wheat
- Fumaria (Active Comparator): Fumaria capsule (0.5 mg Fumaria parviflora L.) / 2 capsule 3 times per day.
  Interventions: Drug: Fumaria

INTERVENTIONS:
Drug: Wheat — 3 times a day each time 2 capsules before eating meal for 8 weeks.
  Arms: Wheat
Drug: Fumaria — 3 times a day each time 2 capsules before eating meal for 8 weeks.
  Arms: Fumaria

SUMMARY:
The purpose of this study is to determine whether Fumaria Parviflora L. can minimize severity of pruritus in patients with end-stage renal disease.

DETAILED DESCRIPTION:
Uremic Pruritus is still a common complication in end-stage renal disease patients. The pathogenesis of Uremic Pruritus is unknown, therefore treatments are ineffective. According to several studies Uremic Pruritus is not an isolated skin disease. It seems to be a systemic inflammatory disease with a deranged balance of T helper cell differentiation. In this study investigators considered to evaluate effect of Fumaria Parviflora L. in uremic pruritus by a double blind placebo control clinical trial. It is hypothesized that oral Fumaria Parviflora L. may minimize uremic pruritus by decreasing serum Interferon gamma (IFN-γ) and high-sensitive C reactive protein (hs-CRP).

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients
* Suffering from pruritus for at least 6 weeks
* Have not responded to other drugs
* visual analogue scale (VAS) equal or more than 4

Exclusion Criteria:

* Liver disease
* Respiratory disease
* Dermatological disease
* Hemoglobin less than 10
* Cholestasis
* Malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Severity of Pruritis as measured by a visual analogue scale (VAS) | 3 months
  A '0' score represented absence of pruritus and a '10' represented the greatest severity of symptoms.

SECONDARY OUTCOMES:
Serum Interferon-gamma level | 4 months
Serum IL-4 level | 4 months
Serum high-sensitive C reactive protein (hs-CRP) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Roozbeh, MD, Study Chair — Shiraz University of Medical Sciences; Pouya Faridi, PhD, Study Director — Shiraz University of Medical Sciences; Rahimeh Akrami, PhD, Principal Investigator — Shiraz University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Fallahzadeh MK, Roozbeh J, Geramizadeh B, Namazi MR. Interleukin-2 serum levels are elevated in patients with uremic pruritus: a novel finding with practical implications. Nephrol Dial Transplant. 2011 Oct;26(10):3338-44. doi: 10.1093/ndt/gfr053. Epub 2011 Mar 3. PMID 21372257
- [Background] Kimmel M, Alscher DM, Dunst R, Braun N, Machleidt C, Kiefer T, Stulten C, van der Kuip H, Pauli-Magnus C, Raub U, Kuhlmann U, Mettang T. The role of micro-inflammation in the pathogenesis of uraemic pruritus in haemodialysis patients. Nephrol Dial Transplant. 2006 Mar;21(3):749-55. doi: 10.1093/ndt/gfi204. Epub 2005 Oct 25. PMID 16249205
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264
- See also: Itching, Kidney Diseases, Kidney Failure — https://www.nlm.nih.gov/medlineplus/
- See also: Fumaria — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp